CLINICAL TRIAL: NCT02731469
Title: Clinical Study of the Pharmacokinetics, Pharmacodynamics, Tolerability, Safety and Immunogenicity of BCD-131 Compared to Mircera and Aranesp in Healthy Volunteers
Brief Title: Study of Pharmacokinetics, Pharmacodynamics, Safety of BCD-131 Compared to Mircera and Aranesp in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BCD-131-1
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2018-10

CONDITIONS: Reticulocyte Count
MeSH Terms: interventions — continuous erythropoietin receptor activator; Darbepoetin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (11):
- BCD-131, 0.05 mcg/kg subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in a dose 0.05 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 0.15 mcg/kg subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in a dose 0.15 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 0.40 mcg/kg subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in a dose 0.40 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 1.05 mcg/kg subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in a dose 1.05 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 1.70 mcg/kg SC (Experimental): Healthy volunteers will receive BCD-131 in a dose 1.70 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 2.25 mcg/kg SC (Experimental): Healthy volunteers will receive BCD-131 in a dose 2.25 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- BCD-131, 4.45 mcg/kg subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in a dose 4.45 mcg/kg subcutaneously
  Interventions: Biological: BCD-131
- Mircera®, 1.20 mcg/kg subcutaneously (Active Comparator): Healthy volunteers will receive Mircera in a dose 1.20 mcg/kg subcutaneously
  Interventions: Biological: Mircera®
- Aranesp®, 0.45 mcg/kg subcutaneously (Active Comparator): Healthy volunteers will receive BCD-131 in a dose 0.45 mcg/kg subcutaneously
  Interventions: Biological: Aranesp®
- BCD-131, optimal dose, intravenously (Experimental): Healthy volunteers will receive BCD-131 in optimal dose determined on first stage of clinical trial intravenously
  Interventions: Biological: BCD-131
- BCD-131, optimal dose, subcutaneously (Experimental): Healthy volunteers will receive BCD-131 in optimal dose determined on first stage of clinical trial subcutaneously
  Interventions: Biological: BCD-131

INTERVENTIONS:
Biological: BCD-131
  Other Names: pegylated darbepoetin alfa
  Arms: BCD-131, 0.05 mcg/kg subcutaneously; BCD-131, 0.15 mcg/kg subcutaneously; BCD-131, 0.40 mcg/kg subcutaneously; BCD-131, 1.05 mcg/kg subcutaneously; BCD-131, 1.70 mcg/kg SC; BCD-131, 2.25 mcg/kg SC; BCD-131, 4.45 mcg/kg subcutaneously; BCD-131, optimal dose, intravenously; BCD-131, optimal dose, subcutaneously
Biological: Mircera®
  Other Names: Methoxy polyethylene glycol-epoetin beta
  Arms: Mircera®, 1.20 mcg/kg subcutaneously
Biological: Aranesp®
  Other Names: darbepoetin alfa
  Arms: Aranesp®, 0.45 mcg/kg subcutaneously

SUMMARY:
BCD-131-1 is an Open-Label Clinical Study of the Pharmacokinetics, Pharmacodynamics, Tolerability, Safety and Immunogenicity of Single Ascending Doses of BCD-131 in Healthy Volunteers

DETAILED DESCRIPTION:
BCD-131 is novel drug product of pegylated darbepoetin alfa.

Clinical trial BCD-131-1 will be conducted in two stages:

Stage I is an open-label, non-randomized clinical study of pharmacokinetics, pharmacodynamics, tolerability, safety and immunogenicity of BCD-131 given to healthy volunteers at ascending doses (Phase 1, a traditional "3+3" design).

Also, the PK and PD parameters of the closest analogues of BCD-131 (Mircera and Aranesp) given as subcutaneous injections at therapeutic doses will be evaluated.

Stage II aims to further evaluate pharmacokinetics, pharmacodynamics and safety of subcutaneous and intravenous injections of BCD-131 at a dose which ensures PD effects similar to those of the closest analogues (Mircera, Aranesp) given as subcutaneous injections at therapeutic doses.

ELIGIBILITY:
Inclusion Criteria:

1. Signing of the Informed Consent Form;
2. Male sex;
3. Age of 18 to 45 years, inclusive;
4. BMI within normal limits (18.5-24.9 kg/m2);
5. Healthy patients, which is proved by their medical history, physical examination and laboratory findings:

   * No clinically significant abnormalities of circulatory, respiratory, nervous, hematopoietic, endocrine and digestive systems, liver and kidneys in the past medical history and at screening;
   * No history of cardiovascular disorders or thyroid disorders;
   * No history of hematologic disorders, including but not limited to any type of anemia, myelodysplastic syndrome, blood cancers, hemolytic syndrome, hemoglobinopathies, coagulopathies;
   * CBC results within normal limits, including:

     * Hemoglobin within 132-173 g/L;
     * Hematocrit (based on CBC results) within 39-49%;
     * Platelet count within 150-400*109/L;
     * Absolute reticulocyte count within 30.4-93.5 * 109/L;
   * Blood biochemistry and urinalysis results within normal limits;
   * Serum ferritin within 20-250 µg/L;
   * Serum endogenous erythropoietin within 4.3-29.0 MIU/mL;
   * Hemodynamic parameters within normal limits: systolic blood pressure within 100-139 mmHg; diastolic blood pressure within 60-90 mmHg; heart rate within 50-90 bpm;
   * No history of chronic infections (tuberculosis) or chronic inflammation;
   * No hepatitis B or C, HIV, or syphilis;
   * No acute infections within 4 weeks prior to inclusion in the study;
   * No psychiatric disorders and other conditions (including depression) that can interfere with the volunteer's ability to follow the study protocol;
   * Well-being (in the volunteer's opinion) within 30 days prior to inclusion in the study;
6. No history of or current (at baseline) alcohol or drug abuse;
7. Ability of the volunteer, in the investigator's opinion, to follow the study protocol procedures;
8. Willingness of volunteers and their sexual partners with preserved reproductive potential to use reliable contraception within 2 weeks before inclusion in the study and up to 7 weeks after the injection of the test product. This criterion is not applicable to subjects who underwent surgical sterilization. Reliable methods of contraception include one barrier method in combination with one of the following methods: spermicides, intrauterine device/oral contraceptives (for sexual partners).
9. Willingness of volunteers to avoid alcohol intake within 24 hours before and 8 days after each injection of the test drug;

Exclusion Criteria:

1. History of treatment with erythropoietins or any other ESAs;
2. Acute bleeding, blood/plasma donation or blood transfusion within 2 months before inclusion in the study;
3. History of chronic bleeding;
4. Standard laboratory and instrumental findings outside normal limits at screening;
5. History of allergies (anaphylactic shock or multiple drug allergy syndrome);
6. Known allergy or intolerance to any components of the investigational product;
7. Major surgery within 30 days prior to screening, or surgery being scheduled for any time during the study;
8. Impossibility to install a venous catheter for blood sampling (e.g. because of skin disorders at the sites of venipuncture);
9. Diseases or other conditions that can interfere with the pharmacokinetics of the investigational drug (e.g. chronic liver, kidney, blood, circulatory system, lung or neuroendocrine diseases, including diabetes mellitus and others);
10. History of fever of 40 °C or more;
11. History of elevated hepatic transaminases (above 2.5xULN);
12. Episodes of thrombosis and/or thromboembolia in past medical history (myocardial infarction, stroke, transient ischemic attacks, deep vein thrombosis, pulmonary embolism within 6 months prior to inclusion in the study) as well as an increased risk of deep vein thrombosis;
13. History of epileptic attacks or seizures;
14. History or current (at screening) depression, suicidal thoughts/ attempts;
15. Regular oral or parenteral use of any medications including over-the-counter drugs, vitamins and nutritional additives within 2 weeks before a scheduled injection of the test drug;
16. Use of drugs, including OTC products, that significantly affect the hemodynamics, hepatic function, etc. (barbiturates, omeprazole, cimetidine, etc.) within 30 days before a scheduled injection of the test drug;
17. Vaccination within 4 weeks before a scheduled injection of the test drug;
18. Smoking more than 10 cigarettes per day;
19. Consumption of more than 10 portions of alcohol per week (one portion equals to 0.5 L of beer, 200 mL of wine or 50 mL of ethanol) or a history of alcohol, drug or medication abuse;
20. Participation in other clinical studies within 1 month before screening or simultaneous participation in another clinical study;
21. Previous participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, PhD, Study Chair — JCS BIOCAD

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-131, 0.05 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 0.05 mcg/kg subcutaneously
  BCD-131
- BCD-131, 0.15 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 0.15 mcg/kg subcutaneously
  BCD-131
- BCD-131, 0.40 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 0.40 mcg/kg subcutaneously
  BCD-131
- BCD-131, 1.05 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 1.05 mcg/kg subcutaneously
  BCD-131
- BCD-131, 1.70 mcg/kg SC: Healthy volunteers received BCD-131 in a dose 1.70 mcg/kg subcutaneously
  BCD-131
- BCD-131, 2.25 mcg/kg SC: Healthy volunteers received BCD-131 in a dose 2.25 mcg/kg subcutaneously
  BCD-131
- BCD-131, 4.45 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 4.45 mcg/kg subcutaneously
  BCD-131
- Mircera®, 1.20 mcg/kg Subcutaneously: Healthy volunteers received Mircera in a dose 1.20 mcg/kg subcutaneously
  Mircera®
- Aranesp®, 0.45 mcg/kg Subcutaneously: Healthy volunteers received BCD-131 in a dose 0.45 mcg/kg subcutaneously
  Aranesp®
- BCD-131, Optimal Dose, Intravenously: Healthy volunteers received BCD-131 in optimal dose - 2,75 mcg/kg determined on first stage of clinical trial intravenously
  BCD-131
- BCD-131, Optimal Dose, Subcutaneously: Healthy volunteers will receive BCD-131 in optimal dose - 2,75 mcg/kgdetermined on first stage of clinical trial subcutaneously
  BCD-131
Period: Overall Study
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Started | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Completed | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 45
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24 [21 to 25] | 26 [22 to 36] | 30 [23 to 40] | 32 [23 to 36] | 26 [26 to 27] | 25 [22 to 32] | 25 [22 to 26] | 28 [22 to 31] | 28 [25 to 31] | 24 [23 to 29] | 25 [25 to 27] | 26 [23 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-1176 Hours)
Description: Area under curve (AUC) "concentration - time" from 0 hours to 1176 hours and to infinity
Time Frame: 0, 15 min, 30 min; 60 min; 2 h, 4 h; 8 h, 24 h, 48 h, 72 h, 96 h, 120 h, 168 h, 216 h, 288 h, 336 h, 504 h, 672 h, 840 h, 1008 h, 1176 h post dose
Measure: Median (Inter-Quartile Range); unit: pg*hr/ml
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
pg*hr/ml | 206974.500 [144988.500 to 485443.500] | 657417.000 [598401.500 to 666088.500] | 827904.750 [362302.000 to 1179816.500] | 1360020.000 [424094.000 to 1427990.750] | 1314197.750 [64430.000 to 1465335.500] | 3202606.500 [2173496.250 to 4300376.000] | 5220198.750 [4658082.250 to 5328878.250] | 688124.000 [478496.000 to 1252376.250] | 94628.375 [49807.250 to 113412.500] | 6382389.188 [4818041.5 to 6826251.75] | 2089193.125 [789943 to 2926898]

2. Secondary Outcome: Cmax
Description: Maximal concentration of drug in blood after single injection
Time Frame: 0, 15 min, 30 min; 60 min; 2 h, 4 h; 8 h, 24 h, 48 h, 72 h, 96 h, 120 h, 168 h, 216 h, 288 h, 336 h, 504 h, 672 h, 840 h, 1008 h, 1176 hours post-dose
Measure: Median (Inter-Quartile Range); unit: picogram per ml
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
picogram per ml | 585.000 [503.000 to 744.000] | 1035.000 [854.000 to 1761.000] | 2248.000 [1457.000 to 2566.000] | 3634.000 [2924.000 to 4954.000] | 3541.000 [150.000 to 4110.000] | 12023.000 [6863.000 to 12243.000] | 15433.000 [13286.000 to 16404.000] | 2298.000 [1849.000 to 6867.000] | 964.500 [870.000 to 1229.000] | 87526.5 [69859 to 93090] | 10588 [3713 to 11692]

3. Secondary Outcome: Tmax
Description: Time from 9 hours to time of maximal concentration of drug in blood after single injection
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
hours | 216.000 [96.000 to 504.000] | 168.000 [72.000 to 504.000] | 96.000 [8.000 to 96.000] | 72.000 [48.000 to 72.000] | 72.000 [48.000 to 168.000] | 120.000 [96.000 to 168.000] | 96.000 [72.000 to 96.000] | 48.000 [48.000 to 72.000] | 36.000 [8.000 to 36.000] | 0.75 [0.5 to 1] | 84 [72 to 96]

4. Secondary Outcome: T1/2
Description: Half-life of drug in blood after single injection. In the coрort BCD-131 0,15 mcg/kg due to the absence of a linear terminal elimination phase in volunteers, the calculation of T1 / 2 was not possible
Time Frame: as for outcome 2
Population: the calculation of the half-life in group 0,15 mcg/kg was not carried out, due to the lack of a linear terminal phase of elimination in volunteers
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 0 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
hours | 322.094 [322.094 to 322.094] |  | 377.272 [281.082 to 473.461] | 212.231 [212.231 to 212.231] | 416.482 [326.648 to 506.316] | 191.477 [145.071 to 495.813] | 181.310 [168.649 to 186.681] | 114.855 [105.888 to 256.031] | 79.473 [44.619 to 104.605] | 116.125 [70.7 to 120.38] | 182.392 [123.71 to 197.76]

5. Secondary Outcome: Kel
Description: Elimination rate constant of drug in blood after single injection. In the cohort BCD-131 0,15 mcg/kg due to the absence of a linear terminal elimination phase in volunteers, the calculation of Kel was not possible
Time Frame: as for outcome 2
Population: the calculation of the Kel in group "0,15 mcg/kg" was not carried out, due to the lack of a linear terminal phase of elimination in volunteers
Measure: Median (Inter-Quartile Range); unit: fraction per hour
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 0 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
fraction per hour | 0.002152 [0.002152 to 0.002152] |  | 0.001965 [0.001464 to 0.002466] | 0.003266 [0.003266 to 0.003266] | 0.001746 [0.001369 to 0.002122] | 0.003620 [0.001398 to 0.004778] | 0.003823 [0.003713 to 0.004110] | 0.006057 [0.003734 to 0.006549] | 0.009019 [0.006697 to 0.019655] | 0.005977 [0.003424 to 0.006196] | 0.003828 [0.001367 to 0.00415]

6. Secondary Outcome: Clearance of BCD-131
Description: Clearance of BCD-131 in blood after single injection
Time Frame: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ml per hour
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
ml per hour | 17.393 [8.446 to 24.140] | 16.200 [15.313 to 21.808] | 33.337 [24.411 to 83.908] | 54.043 [48.530 to 225.304] | 92.812 [91.843 to 1820.580] | 65.259 [46.682 to 88.567] | 51.774 [51.147 to 57.320] | 108.993 [59.886 to 156.741] | 332.263 [304.017 to 602.322] | 29.84 [24.293 to 30.734] | 136.391 [48.481 to 202.399]

7. Secondary Outcome: AUEC (0-1176 Hours) - Reticulocytes
Description: Area under effect curve (AUEC) "absolute reticulocyte count - time" from 0 to 1176 hours post-dose after single injection of study drug
Time Frame: 0, 24 h, 48 h; 72 h; 96 h; 120 h; 168 h; 216 h; 288 h; 336 h, 504 h; 672 h; 840 h; 1008 h; 1176 h post-dose
Measure: Median (Inter-Quartile Range); unit: cells (10^9) * hr/l
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
cells (10^9) * hr/l | 10568.04 [10107.60 to 10940.76] | 348.000 [144.000 to 1980.000] | 2868.000 [2664.000 to 17556.00] | 11004.00 [6006.000 to 13416.00] | 14481.60 [10366.80 to 15530.40] | 25512.00 [16476.00 to 30355.20] | 69120.00 [46183.20 to 81511.20] | 10269.72 [3121.200 to 16310.88] | 14223.60 [8736.000 to 21257.28] | 21370.44 [18081.6 to 22724.88] | 13129.2 [4432.56 to 15072]

8. Secondary Outcome: AUEC (0-1176 Hours) - Hemoglobin
Description: Area under effect curve (AUEC) "hemoglobin - time" from 0 to 1176 hours post-dose after single injection of study drug
Time Frame: 0, 24 h, 48 h; 72 h; 96 h; 120 h; 168 h; 216 h; 288 h; 336 h, 504 h; 672 h; 840 h; 1008 h; 1176 h post-dose
Measure: Median (Inter-Quartile Range); unit: gr*hr/l
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
gr*hr/l | 864.00 [528.00 to 2460.00] | 216.00 [0.00 to 1260.00] | 1992.00 [1152.00 to 3864.00] | 4752.00 [2688.00 to 6924.00] | 1548.00 [1320.00 to 10128.00] | 1392.00 [660.00 to 23460.00] | 3516.00 [2904.00 to 4248.00] | 3492.00 [720.00 to 6156.00] | 3120.00 [2112.00 to 4320.00] | 4008 [2340 to 4044] | 4632 [2448 to 4812]

9. Secondary Outcome: AC-Emax - Reticulocytes
Description: Absolute maximum of reticulocyte count (AC-Emax - reticulocytes) after single injection of study drug
Time Frame: 0, 24 h, 48 h; 72 h; 96 h; 120 h; 168 h; 216 h; 288 h; 336 h, 504 h; 672 h; 840 h; 1008 h; 1176 h post-dose
Measure: Median (Inter-Quartile Range); unit: 10e9 reticulocytes per liter"
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
10e9 reticulocytes per liter" | 23.65 [17.15 to 31.34] | 6.00 [6.00 to 22.00] | 13.00 [11.00 to 34.00] | 27.00 [12.00 to 28.00] | 20.68 [17.00 to 26.00] | 112.00 [81.00 to 132.00] | 110.00 [69.00 to 171.00] | 58.00 [48.00 to 91.42] | 62.22 [48.00 to 153.10] | 70.18 [67 to 72.76] | 57.5 [45.4 to 58]

10. Secondary Outcome: AC-Emax - Hemoglobin
Description: Absolute maximum of hemoglobin (AC-Emax - hemoglobin) after single injection of study drug
Time Frame: 0, 24 h, 48 h; 72 h; 96 h; 120 h; 168 h; 216 h; 288 h; 336 h, 504 h; 672 h; 840 h; 1008 h; 1176 h post-dose
Measure: Median (Inter-Quartile Range); unit: gramm per liter
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
gramm per liter | 8.00 [3.00 to 11.00] | 2.00 [0.00 to 22.00] | 7.00 [5.00 to 9.00] | 9.00 [8.00 to 15.00] | 9.00 [6.00 to 21.00] | 6.00 [4.00 to 26.00] | 10.00 [8.00 to 10.00] | 10.50 [3.00 to 12.00] | 9.00 [8.00 to 13.00] | 11.00 [8.00 to 13.00] | 10.5 [9.00 to 12.00]

11. Secondary Outcome: Intensity of Pain After Subcutaneous Injection According to Visual Analog Scale
Description: visual analog scale Minimum value - 0, Maximum value -10, Higher scores mean worse outcome
Time Frame: intraoperative
Population: In second period of study, when healthy volunteers received BCD-131 in optimal dose, visual analoge scale was not applied (by protocol)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 0 | 0
score on a scale | 0 [0 to 2] | 0 [0 to 0] | 0 [0 to 2] | 2 [0 to 2] | 2 [0 to 2] | 0 [0 to 2] | 2 [0 to 2] | 0 [0 to 0] | 2 [0 to 2] |  |

12. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: Total incidence of adverse events (AE)/ serious adverse events (SAE)
Time Frame: from the first administartion of the drug up to the end of follow up period (28 days after the last dose of the drug)
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 1 | 2 | 2 | 0 | 0 | 2 | 4 | 4 | 4 | 5

13. Secondary Outcome: Number of Participants With Local Reactions
Description: Incidence of administration site reactions
Time Frame: from the first administartion of the drug up to the end of follow up period (28 days after the last dose of the drug)
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With AE/SAE 3-4 Grade CTCAE
Description: Incidence of Grade 3-4 AEs and SAEs.
Time Frame: from the first administartion of the drug up to the end of follow up period (28 days after the last dose of the drug)
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Early Withdrawal Due to AE
Description: Frequency of early withdrawals due to AEs and SAEs
Time Frame: from the first administartion of the drug up to the end of follow up period (28 days after the last dose of the drug)
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Binding Antibodies to BCD-131
Description: Incidence of Binding antibodies to BCD-131 on Day 50 after a single injection of BCD-131
Time Frame: 0, day 50 post-dose
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 3 | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: from the first administration of the first dose of the drug up to the end of follow up period (28 days after the last administration of the drug)
Arm/Group | BCD-131, 0.05 mcg/kg Subcutaneously | BCD-131, 0.15 mcg/kg Subcutaneously | BCD-131, 0.40 mcg/kg Subcutaneously | BCD-131, 1.05 mcg/kg Subcutaneously | BCD-131, 1.70 mcg/kg SC | BCD-131, 2.25 mcg/kg SC | BCD-131, 4.45 mcg/kg Subcutaneously | Mircera®, 1.20 mcg/kg Subcutaneously | Aranesp®, 0.45 mcg/kg Subcutaneously | BCD-131, Optimal Dose, Intravenously | BCD-131, Optimal Dose, Subcutaneously
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/3 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/3 | 1/3 | 2/3 | 2/3 | 0/3 | 0/3 | 2/3 | 4/6 | 4/6 | 4/6 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-131, 0.05 mcg/kg Subcutaneously (N=3) | BCD-131, 0.15 mcg/kg Subcutaneously (N=3) | BCD-131, 0.40 mcg/kg Subcutaneously (N=3) | BCD-131, 1.05 mcg/kg Subcutaneously (N=3) | BCD-131, 1.70 mcg/kg SC (N=3) | BCD-131, 2.25 mcg/kg SC (N=3) | BCD-131, 4.45 mcg/kg Subcutaneously (N=3) | Mircera®, 1.20 mcg/kg Subcutaneously (N=6) | Aranesp®, 0.45 mcg/kg Subcutaneously (N=6) | BCD-131, Optimal Dose, Intravenously (N=6) | BCD-131, Optimal Dose, Subcutaneously (N=6)
platelet count decreased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
monocytes count decreased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
basophils increased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Platelet count increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 2 | 0
AST increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
eosinophils increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0
Neutrophiles decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Leucocytes decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT02731469/Prot_000.pdf
  • Statistical Analysis Plan (2015-09-21): https://cdn.clinicaltrials.gov/large-docs/69/NCT02731469/SAP_001.pdf